CLINICAL TRIAL: NCT02402686
Title: Open-Label, Multi-Center, Non-Interventional Study in Rheumatoid Arthritis (RA) Patients Treated With Tocilizumab SC Monotherapy in Daily Clinical Practice (SIMPACT)
Brief Title: Non-Interventional Study of Tocilizumab Subcutaneous (SC) Monotherapy in Participants With Rheumatoid Arthritis (RA)
Acronym: SIMPACT
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29719
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Tocilizumab for RA in Routine Clinical Practice: Participants from routine clinical practice in Hungary who are receiving treatment for RA with tocilizumab SC according to standard of care and in line with the current summary of product characteristics (SPC)/local labeling and who have no contraindication to tocilizumab therapy as per the local label are eligible for observation.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Dosing and treatment duration of tocilizumab collected as part of this non-interventional study are at the discretion of the physician in accordance with local clinical practice and local labeling. Observation period is 24 weeks from first SC tocilizumab administration.
  Other Names: RoActemra

SUMMARY:
The aim of this non-interventional study in Hungarian participants is to gather real life data about the efficacy and safety of tocilizumab SC monotherapy in RA, to assess data about pattern of usage of tocilizumab monotherapy in RA disease management.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe RA according to 2010 American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR) joint criteria
* Treatment with tocilizumab SC monotherapy for up to 8 weeks prior to enrollment, under the prescriptive authority of a physician who has made the decision to commence tocilizumab in accordance with the local label
* Methotrexate intolerance, or inadequate response to prior DMARDs and TNF inhibitors where continued methotrexate treatment was deemed inappropriate

Exclusion Criteria:

* Treatment with tocilizumab more than 8 weeks prior to enrollment
* Failure to meet local tocilizumab label indication criteria
* Treatment with any investigational agent within 4 weeks of beginning tocilizumab SC monotherapy
* Last methotrexate dose within 1 week of beginning tocilizumab SC monotherapy
* History of any other autoimmune or joint inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants receiving treatment for RA with tocilizumab SC according to standard of care and in line with the current SPC/local labeling and who have no contraindication to tocilizumab therapy as per the local label. This can include participants who have received tocilizumab SC monotherapy treatment within 8 weeks prior to the enrollment visit.
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Change in Disease Activity Score 28 (DAS28) from Baseline to End of Study | Baseline, end of study (up to 24 weeks)

SECONDARY OUTCOMES:
Change in Clinical Disease Activity Index (CDAI) Score from Baseline to End of Study | Baseline, end of study (up to 24 weeks)
Percentage of Participants Achieving DAS28 Remission, as Defined by DAS28 Less Than or Equal to (≤) 2.6 | Up to 24 weeks
Percentage of Participants Achieving CDAI Remission, as Defined by CDAI ≤2.8 | Up to 24 weeks
Change in DAS28 from Baseline to End of Study in Different Monotherapy Subgroups | Baseline, end of study (up to 24 weeks)
  The following 3 monotherapy subgroups will be included: 1) participants starting tocilizumab after failing disease-modifying antirheumatic drugs (DMARDs), 2) participants starting tocilizumab after failing one biologic, 3) participants starting tocilizumab after failing two or more biologics.
Percentage of Participants Achieving DAS28 Remission in Different Monotherapy Subgroups, as Defined by DAS28 ≤2.6 | Up to 24 weeks
  The following 3 monotherapy subgroups will be included: 1) participants starting tocilizumab after failing DMARDs, 2) participants starting tocilizumab after failing one biologic, 3) participants starting tocilizumab after failing two or more biologics.
Number of Tocilizumab SC Injections per Participant During Observational Treatment Period | Up to 24 weeks
Percentage of Participants Who Discontinued Tocilizumab, Categorized by the Reasons for the Discontinuations | Up to 24 weeks
Percentage of Participants on SC Tocilizumab First Line Monotherapy | Up to 24 weeks
Percentage of Participants with Reasons for SC Tocilizumab Monotherapy | Up to 24 weeks
Percentage of Participants Treated Previously with a Tumor Necrosis Factor (TNF) Inhibitor/Other Biologic and Low Dose Methotrexate (Less Than 10 Milligrams/Week) | Up to 24 weeks
Percentage of Participants with Other DMARDs Than Methotrexate Before Tocilizumab Monotherapy Initiation and at End of Observation Period | Baseline, Week 24
Percentage of Participants with Oral Steroid at Initiation of Tocilizumab SC Therapy and at End of Study | Baseline, Week 24
Percentage of Participants With Steroid Dose Reductions/Withdrawal at End of Observation Period | Week 24
Percentage of Participants with Steroid Tapering in Different Monotherapy Subgroups Who Achieved DAS28 Remission | Up to 24 weeks
  The following 3 monotherapy subgroups will be included: 1) participants starting tocilizumab after failing DMARDs, 2) participants starting tocilizumab after failing one biologic, 3) participants starting tocilizumab after failing two or more biologics.
Percentage of Participants with Adverse Events | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- Hungary (18):
  - National Institute of Rheumatology and Physiotherapy; 4Th Rheumatology Department, Budapest
  - Budai Irgalmasrendi Kórház KHT. II. Reumatológia, Budapest
  - Magyar Honvedseg Honved Korhaz, Reumatologia, Budapest
  - Debreceni Egyetem Orvos- és Egészségtudományi Centrum; Belgyógyászati Intézet, Reumatológiai Tanszék, Debrecen
  - Markhot Ferenc Hospital; Dep. of Rheumatology, Eger
  - Vaszary Kolos Kórház, Esztergom
  - Petz Aladár County Teaching Hospital, Győr
  - Pandy Kalman Hospital; Dept. of Infectious Diseases, Gyula
  - Szent Andras Reumakorhaz; Reumatologia, Hévíz
  - Bacs-Kiskun Megyei Korhaz, Kecskemét
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Szent Ferenc Kórház; Reumatológia, Miskolc
  - Szabolcs-Szatmar-Bereg Megyei Josa Andras Korhaz; Reumatologia, Nyíregyháza
  - Pécsi Tudományegyetem Klinikai Központ: Immunológiai és Reumatológiai Klinika, Pécs
  - Szegedi Tudomanyegyetem Aok Szent-Gyorgyi Albert Klinikai Kozpont; Rheumatologiai Klinika, Szeged
  - Fejér Megyei Szent György Kórház; Reumatológiai Osztály, Székesfehérvár
  - Markusovszky Hospital, Szombathely
  - Veszprém Megyei Csolnoky Ferenc Kórház; Reumatológia, Veszprém

REFERENCES:
- [Derived] Nagy G, Geher P, Tamasi L, Drescher E, Keszthelyi P, Pulai J, Czirjak L, Szekanecz Z, Kiss G, Kovacs L. Real-world evidence on methotrexate-free subcutaneous tocilizumab therapy in patients with rheumatoid arthritis: 24-week data from the SIMPACT study. Rheumatol Adv Pract. 2022 May 16;6(2):rkac038. doi: 10.1093/rap/rkac038. eCollection 2022. PMID 35663154